CLINICAL TRIAL: NCT05116319
Title: Sensitivity and Specificity of Guidelines' Recommendations and Existing Predictive Models to Detect Undiagnosed Diabetes Mellitus or Prediabetes in a Chinese Population
Brief Title: Prediction to Detect Pre-DM/DM in a Chinese Population
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CREC-202103
Record Dates: First submitted 2021-10-20; First posted 2021-11-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese people with no known history of diabetes
  Interventions: Diagnostic Test: point-of-care HbA1c

INTERVENTIONS:
Diagnostic Test: point-of-care HbA1c — The Afinion2™ (Abbott, Oslo, Norway), will be used for the current study as it is recently validated. According to American Diabetes Association (ADA), pre-diabetes (pre-DM) is diagnosed if HbA1c is 5.7-6.4% and diabetes (DM) is diagnosed if HbA1c is ≥6.5%

SUMMARY:
This project will compare the sensitivity and specificity of different screening criteria or recommendations to detect pre-diabetes or diabetes mellitus in a Chinese population, using point-of-care hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* age ≥25 years old
* with no previous diagnosis of DM
* Chinese.

Exclusion Criteria:

* a history of cardiovascular diseases including any type of stroke, ischemic heart disease, atrial fibrillation, and/or peripheral vascular disease
* severe mental or physical disease or language barriers that limited data collection

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Chinese population
Sampling Method: Non-Probability Sample
Enrollment: 1901 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Point-of-care (POC) HbA1c | baseline
  the measurement to diagnose pre-diabetes or diabetes; pre-DM is diagnosed if HbA1c is 5.7-6.4% and DM is diagnosed if HbA1c is ≥6.5%.

SECONDARY OUTCOMES:
Office blood pressure | baseline
  a measurement to screen for hypertension; BP will be measured for 2 times (1-minute apart) and will be in accordance to the Hong Kong Primary Care Office guideline (e.g. the choice of cuffs and positioning). The average of the two BP readings will be used for analysis and management. Elevated BP is defined as a systolic BP (SBP) of ≥140mmHg and/or a diastolic BP (DBP) ≥90mmHg
Body mass index | baseline
  a measurement for obesity. Body mass index (BMI) is calculated by weight divided by the square of height (BMI = weight (kg)/height(m)2). According the Hong Kong Centre for Health Protection, overweight and obesity are defined as a BMI of 23-24.9kg/m2 and ≥25kg/m2 respectively

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Will share data upon researchers' reasonable request